CLINICAL TRIAL: NCT00274170
Title: Randomized Evaluation of Octreotide Versus Compazine for Emergency Department Treatment of Migraine Headache
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2006.014
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Migraine Headache
Keywords: Migraine; Octreotide; Prochlorperazine
MeSH Terms: conditions — Migraine Disorders | interventions — Octreotide

INTERVENTIONS:
Drug: Octreotide

SUMMARY:
: Headaches are a common complaint presenting to the emergency department (ED), accounting for 1-2% of all ED visits, with migraines as the second most common primary headache syndrome. Patients that ultimately present to the ED have failed outpatient therapy and exhibit severe and persistent symptoms. Treatment options have been traditionally with a parenteral opiod, generally Demerol. Unfortunately, patients with chronic painful conditions like migraines have been prone to dependency. In 1986, a nonopioid, compazine was noted serendipitously to relieve migraine headache pain. 1 Nonopioid regimens have evolved as standard therapy in the treatment of migrainne headache in the ED. Today, there are a number of nonopioid treatment options, but not without their own individual concerns. Ergotamine and dihydroergotamine are effective, but commonly cause nausea and vomiting. Sumatriptan is expensive has recurrence rate, is ineffective in about 20-30%, and is contra-indicated in patients with cardiac disease. Metoclopramide, a dopamine receptor antagonist, commonly used as an anti-emetic agent, has been widely studied for use with acute migraines. Its side effects include drowsiness and dystonic reactions. Compazine has been successfully used to treat migraine headaches for the past several decades, and has been accepted as standard treatment of headaches in the ED. 2 Its side effect profile includes extrapyramidal effects, dysphoria, drowsiness and akathisias. The ideal medication for treating headaches would have no addictive properties, few side effects, quick onset, be highly effective and have a low rate of recurrence. Somatostatin is known to have an inhibitory effect on a number of neuropetides, which have been implicated in migraine. Native somatostatin is an unstable compound and is broken down in minutes, but octreotide, a somatostatin analogue has a longer half life. Intravenous somatostatin has been shown to be as effective as ergotamine in the acute treatment of cluster headache. 3 The analgesic effect of octreotide with headaches associated with growth hormone secreting tumor has been established. 4 Five somatostatin receptors have been cloned with octreotide acting predominantely on sst2 and sst5. The distribution of sst2 within the central nervous system strongly suggests that this particular somatostatin receptor has a role in cranial nociception, being highly expressed in the trigeminal nucleus caudalis and periaqueductal grey. Kapicioglu et.al performed a double blind study comparing octreotide to placebo in treating migraine. They found there to be a significantly greater relief of pain with octreotide at 2 and 6 hours compared to placebo (76% vs 25%, p<0.02). They noted that 47% of those in the octreotide group had complete relief compared to no patients in the placebo group. They went on to note that those patients in the octreotide group had earlier relief of symptoms and no side effects. The only minor adverse event related to the administration of octreotide was a local reaction in 3 patients (18%). In a study performed recently in Netherlands, no clinically relevant changes in vital signs, routine chemistry, and urinalysis were observed with octreotide use. Electrocardiogram analyses showed no newly occurring or worsening of known cardiac abnormalities 2 and 24 h after injection with octreotide. 5 Levy et. al also compared octreotide to placebo in a double blinded study but found no difference. This was a poorly designed study, in that the patients treated themselves at home with an injection of either placebo or octreotide for 2 episodes of headache and recorded their level of pain relief at 2 hours. Matharu et. al also performed a double blind study comparing octreotide to placebo, but looking at cluster headaches rather than migraines. They found there to be a significant improvement with the use of octreotide over placebo (52% vs 36%). At Darnall Army Community Hospital the cost of 100 mcg Octreotide and10 mg Compazine, is $10.46, $2.02-8.00, respectively.

DETAILED DESCRIPTION:
A urine pregnancy test will be performed on women of child bearing age. After informed consent is obtained, each patient will be placed in a dark private room and asked to grade nausea, pain, and sedation on a 10 cm visual analog scale, using the left end as the zero point for complaints and measurements. Patients will be instructed that a score of zero signifies no pain and a score of 10 indicates severe pain. Each patient will be monitored with continous pulse oximetry and have a 20-gauge IV catheter placed in the antecubital fossa. Based on a computer generated random table, each subject will receive one of the following: 2 cc containing 100ug octreotide, or 10 mg compazine over a 2 minute period, followed by a 5 cc flush of saline solution. The above medication doses were chosen based on previous literature. 6-8 Vital signs (blood pressure, heart rate, and respiratory rate) will be recorded at 0, 30, and 60 minutes. At 60 minutes after the study injection, each patient will be asked to regrade nausea, pain(VAS), and sedation on the same scale without viewing the initial scores. Clinically important successful treatment will be defined as achievement of the following criteria: patient satisfaction and either a decrease of 50% or more in the pain score (compared with the initial score) or an absolute pain score of 2.5 cm or less. Failure to achieve these criteria constitute treatment failure. The treating physician will use an acceptable rescue medicine or group of medicines at treatment failure. The 60 minute outcome was selected because of the route chosen (maximal absorption and distribution within minutes) and because previous published data suggests that most responders are identified during this interval. 9 Each patient will be contacted within 48 hours of discharge to define early relapse rate.

4.8 Inclusion criteria: Adults between the age of 18 and 65 years of age and diagnosis of migraine with or without an aura who met the criteria of the International Headache Society, and with at least one prior episode of a similar headache. 10 The International Headache Society diagnosis criteria for migraine with and without aura is outlined in the below table:

Migraine with AuraØ At least two attacks fulfilling the below characteristicsØ Headache has at least three of the following four characteristics:1. 0ne or more fully reversible aura symptoms indicating focal cerebral cortical and/or brain stem dysfunction2. At least one aura symptom develops gradually over more than 4 minutes, or tow or more symptoms occur in succession3. No aura symptom lasts more than 60 minutes; if more than one aura symptom is present, accepted duration is proportionally increased4. Headache follows aura with a free interval of less than 60 minutes (it may also begin before or simultaneously with the aura) Migraine without AuraØ At least 5 attacks fulfilling the below characteristicsØ Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)Ø Headache has at least two of the following four characteristics:1. Unilateral location 2. Pulsating quality 3. Moderate or severe intensity which inhibits or prohibits daily activities 4. Aggravated by walking stairs or similar routine physical activityØ During headache at least one of the two following symptoms occur:1. Nausea and/or vomiting2. Photophobia and phonophobia

4.9 Exclusion criteria: pregnancy and lactation, pre-medication within six hours of being enrolled in the study, more than six prior headaches per month, allergy to the study drugs, non-migraine headache, substance abuse, alcohol abuse, diabetes mellitus, or a coexisting condition that might expose the patients to a disproportionately increased risk of a significant adverse event: ischaemic heart disease, peripheral vascular disease, cerebrovascular disease, uncontrolled hypertension (blood pressure >160/95), epilepsy, use of cimetidine, dopamine agonist, cyclopsorin, or oral hypoglycemic agents, hepatic or renal failure, and thyroid disorder.

4.10 Number of Subjects: TOTAL NUMBER OF SUBJECTS (nation-wide/study-wide) 56

5.0 Human Subject Protection

5.1 Recruitment: Patients presenting to the DACH ER with a complaint of headache will interviewed by the physician. If they meet the inclusion and exclusion criteria, they will be informed about the study by the treating physician, have to opportunity to ask questions, and read the consent form.

5.2 Benefits: Patients participating in this study will have the potential benefit of having their headache pain resolved. They will be part of an effort to find a treatment for migraine headaches that will hopefully be effective and with a lower side effect profile.

5.3 Risks: The risks of this study include treatment failure and an allergic reaction to one of the study medicines. Each medicine cares its own specific risk to the patient due to its unique make-up and mechanism of action.

Octreotide has been shown to inhibit gallbladder contractility and decrease bile secretion in normal volunteers. In clinical trials, the incidence of biliary tract abnormalities was 63% (27% gallstones, 24% sludge without stones, 12% biliary duct dilatation). Less than 2% of patients treated with octreotide for 1 month or less developed gallstones. Octreotide alters the balance between the counter-regulatory hormones, insulin, glucagon and growth hormone, which may result in hypoglycemia (3%) or hyperglycemia (16%). Studies have also demonstrated that octreotide suppress thyroid stimulating hormone (12%). Pancreatitis, bradycardia, poor dietary fat and B12 absorption have also been reported. Most reports are in patients with acromegaly who are prone to the before mentioned problems and the true incidence in the non-acromegaly population is not known.

Compazine has been shown to cause orthostatic hypotension and extrapyramidal symptoms. Of the extrapyramidal symptoms, akathisia (25-60% after single dose) and dystonic reactions (4% after single dose) are the most commonly encountered. These reactions can be minimized by the rate of administration and the concurrent use of diphenhydramine. Due to the study design, diphenhydramine will not be used but a slow rate of administration with 50 ml normal saline bag that will be given over 5 minutes. This slower rate of administration will decrease risk of extrapyramidal symptoms. Irreversible tardive dyskinesia and neuroleptic malignant syndrome have been described with compazine. These complications are extremely rare and the true incidence is unknown

5.4 Safeguards for Protecting Subjects: Data collection sheets will be available to the treating physician and PI only. The PI and AIs will obtain the follow up information for all participants. Adverse reaction to any of the medications will be managed in the emergency department depending on the specific reaction.

5.5 Risk:Benefit Assessment: The medications used in this study are currently being used to treat headaches. Octreotide has been studied in this setting and side effect profile has been minimal. The risks are minimal with the current exclusion criteria. Benefit of relief of headache outweighed the risk of the side effects of any one of these medications.

5.6 Alternatives: Other medications have been used to treat migraines to include morphine, reglan, magnesium. Alternative is also to not to participate in this study.

6.0 Data Analysis: In this study, the independent variables are treatment (octreotide, comparzine, demerol) and time (0, 30, 60 minutes). The dependent variable is pain measured on a numerical rating scale (1 to 10). The null hypothesis is that there will be no difference in pain between treatments. The alternative hypothesis is that there will be a greater decrease in pain with octreotide. The investigator expects the pain at baseline to be 6 +/- 2. A 30% difference in pain between treatments will be clinically significant. This is a 0.3 * 6 / 2 = 0.9 effect size. The appropriate test is a two-factor ANOVA (treatment, time) with repeated measures on one factor (time) followed by one-tailed t-tests corrected for multiple comparisons. Six post hoc comparisons on a one-tailed test are appropriate for this design, so we made a maximum Bonferroni correction of p = 0.05 / 6 = 0.0083 ~ 0.005. I used a look-up table based on employing the method of Kraemer and Thiemann (1988) to obtain an initial estimate of the sample size, which was confirmed with 1000 iterations of a Monte Carlo simulation until the power was between 80% and 85% with a level of confidence of 95%. According to this method, a sample size of 32 per group (96 total) is needed to detect a clinically significant difference with the desired level of confidence and power. If two treatments (octreotide, comparzine) are used, a sample size of 28 per group (56 total) is needed.

ELIGIBILITY:
Inclusion Criteria:

* Migraine Headache

Exclusion Criteria:

* Pregnancy and lactation,
* Pre-medication within six hours of being enrolled in the study,
* More than six prior headaches per month,
* Allergy to the study drugs,
* Non-migraine headache,
* Substance abuse,
* Alcohol abuse,
* Diabetes mellitus, or a coexisting condition that might expose the patients to a disproportionately increased risk of a significant adverse event: ischaemic heart disease, peripheral vascular disease, cerebrovascular disease, uncontrolled hypertension (blood pressure >160/95), epilepsy, use of cimetidine, dopamine agonist, cyclopsorin, or oral hypoglycemic agents, hepatic or renal failure, and thyroid disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2006-01; Study Completion 2007-02

PRIMARY OUTCOMES:
Patient Satisfaction
Improvement of Pain
Improvement of Nausea

CONTACTS AND LOCATIONS:
Overall Officials: Alex Rosin, MD, Principal Investigator — C.R.Darnall Army Medical Center
Locations (1):
- CR Darnall Army Medical Center, Fort Hood, Texas, United States